CLINICAL TRIAL: NCT06631950
Title: A Video Intervention on Young Adults' Fertility Awareness: a Large-scale Educational RCT in Denmark and Norway Measuring Fecundity Knowledge, Fertility Intentions, Reproductive Behavior and Long-run Impacts on Realized Fertility
Brief Title: Young Adults' Fecundity Knowledge and Fertility Intentions and Reproductive Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish National Birth Cohort (DNBC) (Unknown); Norwegian Mother and Child Cohort Study (MoBa) (Unknown); ERC Synergy Grant (European Union, 101071773) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIOSFER RCT - 101071773
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: The Focus is to Investigate Effect of an Educational Video on Fecundity Knowledge Among Young Adults
Keywords: Fecundity knowledge; Fertility awareness; Family intentions; Video intervention
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fecundity knowledge intervention (Experimental): In the experimental arm, participants receive a short (3 minutes) educational video on risk factors of importance for fecundity.
  Interventions: Other: Educational intervention
- Control (No Intervention): In the no-intervention arm, the participants do not receive the intervention (a short educational video).

INTERVENTIONS:
Other: Educational intervention — The educational intervention group will be provided with information that should allow them to correctly answer questions on fecundity knowledge and fecundity risks factors. The fecundity information will be provided through a short animated educational video (3 minutes) that will be sent out digitally. The control group is not receiving such information.
  Arms: Fecundity knowledge intervention

SUMMARY:
This RCT investigates the impact of an educational video on fecundity knowledge among young adults. The video discusses several risk factors associated with fecundity, such as age and smoking. The primary outcome measure of the RCT is fecundity knowledge. The knowledge level is defined based on the following factors: Age; smoking; sexually transmitted infections; Success of spontaneous pregnancy according to female age; Success of pregnancy according to female age and fertility treatment. The secondary outcomes are: intentions regarding the timing of desired pregnancy/childbirth; fecundity-protective behaviors; life goals; realized fertility later in life.

DETAILED DESCRIPTION:
This study is an experimental randomized controlled trial (RCT) based on data from the Danish National Birth Cohort (DNBC) and the Norwegian Mother and Child Cohort Study (MoBa). The RCT consists of young adult offspring from these two birth cohorts. The participants in the subsample will randomly be assigned to either an intervention or a control group. The RCT is part of the research project BIOSFER which is funded by an ERC Synergy Grant (European Union, 101071773). The research project aims to investigate the biologic and social causes of low fertility in modern societies.

The Danish National Birth Cohort (DNBC) is an ongoing nationwide cohort of women and their children with more than 20 years of follow-up data (Olsen et al., 2001). The cohort contains 92,000 women recruited 1996 to 2002, who experienced 100,000 pregnancies in total. It has a rich set of background variables including child's development and health up to 18 years, as well as self-reported measures from age 18 onwards. The oldest offspring in the DNBC will be 29 years old at the time of treatment.

The Norwegian Mother, Father and Child Cohort Study (MoBa) is built around 110,000 pregnancies recruited between 1999 and 2008 (Magnus et al., 2016). Children have reported on their own health and exposures from the age of 13, and health and socioeconomic status were reported by the parents before this age. The RCT study will be conducted on a subsample of the MoBa children who are at least 18 years old as of 2024. The oldest offspring in the MoBa will be 25 years old at the time of treatment.

Data collection for the RCT will take place between late 2024 and mid-2025. The RCT intervention group will receive a fecundity knowledge intervention. The intervention consists of a short (3 minutes) animated educational video containing information on risk factors of importance for fecundity.

The primary outcome measure of the RCT is fecundity knowledge. The knowledge level is defined based on the following factors: Age; smoking; sexually transmitted infections; Success of spontaneous pregnancy according to female age; Success of pregnancy according to female age and fertility treatment. The secondary outcomes are: intentions regarding the timing of desired pregnancy/childbirth; fecundity-protective behaviors; life goals; future reproductive behavior- including attempts to conceive, termination of pregnancies and realized fertility The primary and secondary outcomes are measured with validated self-reported questionnaire items - except for certain items under reproductive behavior, such as 'realized fertility', which is measured through registries.

The target group is adult offspring of the two cohorts, the DNBC and MoBa. Outcomes of the trial will be analyzed for the total population participating in the RCT; for specific age-groups; for men and women; by socioeconomic status of the individuals and their families or origin; and for individuals with high and low risk preferences (measured through questionnaires).

Hypothesis: young adult women and men have low-moderate fecundity knowledge and an educational digital intervention will have an impact on the interventions' group fecundity knowledge and influence a) their family building intentions to desire a first and/or last child at a younger age, b) their fecundity-protective behaviors, c) their priority of life goals, d) their future reproductive behavior, including attempts to conceive, termination of pregnancies and realized fertility.

The goal is to enhance young adults' fecundity knowledge in order to secure that adults are able to make well-informed decisions regarding their family building and reproductive choices.

Individuals who are included in the RCT sample, will be randomized 1:1 by simple randomization to one of the following study arms:

I. Experimental arm (fecundity knowledge intervention group). In the experimental arm, Individuals receive a short (3 minutes) animated educational video on risk factors of importance for fecundity.

II. Control arm (no fecundity knowledge provided).

The investigators will use computer-based randomization methods. When analyzing the data, the data set will by necessity contain information on whether each individual is in the intervention or control group. Coding and classification of outcome variables will be done jointly for the intervention and control group, so this knowledge will not influence the investigators handling of the data.

The intervention group will be provided with information that should allow them to correctly answer questions on fecundity knowledge and fecundity risks factors. The fecundity information will be provided through a short animated educational video that will be sent out digitally. The control group is not receiving such information. As part of the overall BIOSFER project, all offspring in both birth cohorts have received a Global Questionnaire at baseline including items and scales measuring fecundity knowledge and the participants' family formation/intentions regarding family formation and views on life goals. Only participants' having responded to the Global Questionnaire will be invited to the RCT study. After the intervention, both the intervention and the control group will receive identical questionnaire items and scales on fecundity knowledge and intentions regarding family formation, and their views on life goals. Hence, all the respondents receive the questions that inform our outcome variables both before and after the intervention. The participants in the intervention and control group will also be asked about their fecundity-protective behavior.

Statistical analysis and interpretation of data:

Overall, 13,106 (23%) of MoBa participants have responded to the Global Questionnaire. In DNBC data collection of the Global Questionnaire will continue until April 2025. Currently, 11,900 (27% of those who has been invited so far) have responded to the Global Questionnaire. Participants responding to the Global Questionnaire in DNBC and MoBa will receive an invitation to the RCT study.

For the sample size calculation for the primary outcome the investigators expect a participation of 30%. This is based on previous response rates within similar data collections in the two cohorts. Power calculations for the primary outcome were performed with a 5% significance level. The investigators follow convention and use 80% power as a cutoff for sufficient power. Assuming a response rate of 30, there will be power to detect effects down to 5 percent (2.5pp) in the full sample, and 10 percent (5 pp) among women and men when analyzed separately.

The investigators also performed power calculations assessing how power varies as a function of sample size and effect size. The MoBa cohort is used as example, where the RCT invitation will be sent to all 13 106 respondents of the MoBa Global Questionnaire. The investigators also assess the power for sex-specific analysis, with 8325 women and 4723 men (58 answering "other" are excluded from these). The power calculation assumes an even split between groups, and then tests the power for difference in means.

In the power calculations, the investigators use a "fertility knowledge percentage correct score" (see e.g. Bunting et al 2013), with a range from 0 to 100%. The investigators assume a baseline of knowledge of 50 percentage points, somewhat less than what was found in Bunting et al. 2013 (65-68 points). The investigators expect the knowledge level to be lower in our population compared to the population in Bunting et al. 2013. The population in this study is younger (18-29) compared to Bunting et al.'s (31.8 years old). Further, 26% of Bunting et al.'s population already had children, which is expected to be lower in our population. Hence, younger age and not being a parent will most likely effect the knowledge level. With a standard deviation of 25 (taken from Bunting et al. 2013 p. 389), the investigators then assess the power to detect effects of 2.5, 5, 7.5 and 10 percentage points.

Across all samples and down to a 10% response rate, the investigators can detect effects of 7.5 percentage points or higher. In the combined sample, the investigators can detect effects as small as 5 percentage points at a 10% response rate. To detect the smallest effects (2.5 percentage points), a 30% response rate is required for the combined sample.

For women, the investigators can detect effects as small as 5 percentage points with a 10% response rate. To detect effects of 2.5 percentage points require a 40% response rate. In the male sample, effects of 7.5 percentage points and larger can be detected with a 10% response rate. Detecting a 5 pp effect requires 20% response, and 2.5 pp requires more than 50% response.

The effectiveness of the RCT will be analyzed using an intention-to-treat (ITT) approach.

The results of the quantitative evaluation (primary and secondary outcomes) is planned to be analyzed and published in more than one scientific paper.

The quantitative evaluation of RCT is complemented by a qualitative evaluation looking into the participants' thoughts on the fecundity knowledge intervention, highlighting what works for whom under which circumstances, but also their overall thought on family formation.

ELIGIBILITY:
Inclusion Criteria:

* Offspring of mothers part of the DNBC and MoBa cohorts
* Being of legal age
* Responded to the Global Questionnaire at baseline

Exclusion Criteria:

* Being underage
* Not understanding Norwegian/Danish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2045-10 (Estimated)

PRIMARY OUTCOMES:
Change in fecundity knowledge | Measured immediately after intervention (educational video), and at a later point of time (likely within 1-2 years) depending on the data collection logistics for the two cohorts
  Fecundity knowledge level in intervention arm versus control arm. Fecundity knowledge is measured with validated self-reported questionnaire items; revised Cardiff Fertility Knowledge Scale. The values range from 1-100, higher scores indicate higher knowledge level.
  The knowledge level is defined as change in knowledge level of the following factors:
  * Age, smoking, STI (Chlamydia)
  * Success of spontaneous pregnancy according to female age
  * Success of pregnancy according to female age and fertility treatment

SECONDARY OUTCOMES:
Change in intentions regarding timing of pregnancy/childbirth | Measured immediately after intervention (educational video), and at a later point of time (likely within 1-2 years) depending on the data collection logistics for the two cohorts
  Preferred age at first and last child in intervention group compared to the control group. Measured with self-reported questionnaire items.
  Probability of intending to have a child in the near future (1-2 years), and in the relatively near future (up to 4-5 years)
Change in life goals | Measured immediately after intervention (educational video), and at a later point of time (likely within 1-2 years) depending on the data collection logistics for the two cohorts
  Life goals in the intervention group, compared to the control group, are shifted toward emphasis on childbearing and union formation relative to other life goals. Measured with self-reported questionnaire items.
Change in adopting fecundity-protective behaviors | Measured immediately after intervention (educational video), and at a later point of time (likely within 1-2 years) depending on the data collection logistics for the two cohorts
  Intentions of adoption fecundity-protective behaviors in the intervention group compared to the control group. Measured with self-reported questionnaire items.
Change in realized fertility (followed up in registers) | 3, 5, 10 years and 20 years follow-up in national birth registers' after the intervention.
  Total number of children in the intervention group compared to the control group. Followed up in national birth registers' after the intervention.
Change in realized fertility (followed up in registers) | 3, 5, 10 years and 20 years follow-up in national birth registers' after the intervention.
  Mean age at first and at last child in the intervention group compared to the control group. Followed up in national birth registers' after the intervention.
Change in realized fertility (followed up in registers) | 3, 5, 10 years and 20 years follow-up in national birth registers' after the intervention.
  Total number of pregnancy terminations in the intervention group compared to the control group. Followed up in national birth registers' after the intervention.
Change in realized fertility (followed up in registers) | 3, 5, 10 years and 20 years follow-up in national birth registers' after the intervention.
  Mean age at first and at last pregnancy termination in the intervention group compared to the control group. Followed up in national birth registers' after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Myrskylä, Professor, Principal Investigator — Max Planck Institute for Demographic Research, Rostock, Germany; Cecilia Ramlau-Hansen, Professor, Principal Investigator — Department of Public Health - Department of Epidemiology, Aarhus University, Denmark; Siri Eldevik Håberg, Professor, Principal Investigator — Centre for Fertility and Health, Norwegian Institute of Public Health, Norway
Locations (2):
- Aarhus University/DNBC/SSI, Aarhus, Denmark
- Norwegian Institute of Public Health/MoBa, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
For data access, parties must contact DNBC and/or MoBa directly. The new research project must be approved by Danish or/and the Norwegian authorities and follow the procedures for data access in the DNBC/MoBa. All costs for assessing data will be covered by the party requesting the data.